CLINICAL TRIAL: NCT04402099
Title: Study KBP-2020-CPHG Documenting New Cases of Primary Lung Cancer (PLC) Diagnosed in Respiratory Medicine Departments and Lung Cancer Units at General Hospitals From January 1st to December 31st 2020
Acronym: KBP-2020-CPHG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Collège des Pneumologues des Hôpitaux Généraux (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A00943-54
Record Dates: First submitted 2020-04-27; First posted 2020-05-26 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Twenty years after KBP-2000-CPHG study and ten years after KBP-2010-CPHG study, the CPHG proposes to conduct a new epidemiological study on primary PLC in order to evaluate and analyze the changes that have occurred over the last decade.

Primary endpoint:

Estimate 1-year- and 5-year-mortality rates in patients with PLC.

Secondary endpoints:

* Describe PLC patient population managed by pulmonologists at French General Hospitals in 2020
* Describe PLC diagnostic and therapeutic management by pulmonologists at French General Hospitals in 2020 and compare them to KBP-2000-CPHG and KBP-2010-CPHG studies
* Estimate prognostic factors
* Compare patient and tumor characteristics to those observed for KBP-2010-CPHG and KBP-2000-CPHG studies
* Compare observed survival rates to those reported for KBP-2000-CPHG and KBP-2010-CPHG studies

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Primary Lung Cancer histologically (or cytologically or presence of a mutation on liquid biopsy with compatible imaging) proven between January 1st and December 31st, 2020*
* Follow-up by a lung specialist at a General Hospital
* Oral informed consent * date of collected sample

Exclusion Criteria:

* Age < 18 years
* Secondary lung cancer
* Recurrence of same histological type PLC- left to the investigator discretion according to the clinic and the imagery
* Previous enrolment in the study
* Freedom deprived patient following a legal or administrative decision
* Patient unable to give his(her) consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary Lung Cancer histologically proven between January 1st and December 31st, 2020
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Estimate 1-year mortality rates in patients with PLC. | 1 year
  Global survival at 1 year
Estimate 5-year mortality rates in patients with PLC. | 5 years
  Global survival at 5 years

SECONDARY OUTCOMES:
Describe PLC patient population managed by pulmonologists at French General Hospitals in 2020 | 1 year
  - Patient data: age, gender, birth location, height, weight, comorbidity score, smoking status, cannabis uptake, Performance Status, and death
Describe PLC diagnostic and therapeutic management by pulmonologists at French General Hospitals in 2020 and compare them to KBP-2000-CPHG and KBP-2010-CPHG studies | 1 year
  - Disease data: diagnostic method, anatomopathological classification, PDL-1 status, molecular biology test, tumor mutation burden, TNM classification, and stage (8th edition)

CONTACTS AND LOCATIONS:
Locations (1):
- Collège des Pneumologues des Hôpitaux Généraux (CPHG) (General Hospital Pulmonologists College), Paris, France

REFERENCES:
- [Derived] Debieuvre D, Falchero L, Molinier O, Couraud S, Cortot A, Meyer N, Asselain B, Auvray E, Templement-Grangerat D, Bizieux A, Tredaniel J, Schneider S, Auliac JB, Bylicki O, Letierce A, Morel H. Survival of Patients with Lung Adenocarcinoma Diagnosed in 2000, 2010, and 2020. NEJM Evid. 2025 Jul;4(7):EVIDoa2400443. doi: 10.1056/EVIDoa2400443. Epub 2025 Jun 24. PMID 40552964